CLINICAL TRIAL: NCT03047525
Title: The Opening and Negative Controlled Clinical Study of Autologous Multiple Targets DC-CTL Combined With CIK for Advanced Solid Tumor
Brief Title: Study of DC-CTL Combined With CIK for Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaoyi Huang (Other)
Responsible Party: Sponsor-Investigator, Xiaoyi Huang, Director of The Heilongjiang Cancer Biotherapy Center, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMU-2016-002
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Colorectal Cancer; Renal Cell Carcinoma; Nasopharyngeal Carcinoma; Lung Cancer
Keywords: cytokine-induced killer cell; dendritic and cytokine-induced killer cells
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Renal Cell; Nasopharyngeal Carcinoma; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): patients will just regularly chemotherapy
- DC-CIK and CIK Immunotherapy (Experimental): patients will receive chemotherapy with 4 cycles of DC-CIK treatment and 4 cycles of CIK treatment .
  Interventions: Biological: Cytokine-induced Killer Cells

INTERVENTIONS:
Biological: Cytokine-induced Killer Cells — Concurrent of chemotherapy plus 4 cycles of Dendritic and Cytokine-induced Killer Cells(DC-CIK) treatment and 4 cycles of Cytokine-induced Killer Cells(CIK) treatment
  Other Names: DC-CIK and CIK
  Arms: DC-CIK and CIK Immunotherapy

SUMMARY:
Background: Combinations of Dendritic and Cytokine-induced Killer Cells (DC-CIK) and Cytokine-induced Killer Cells (CIK) treatment may enhance the immune response and stop cancer cells from growing. The investigators suppose that DC-CIK combined with CIK treatment will improve the prognosis of advanced solid tumors.

Objective: Phase II clinical trial to investigate the efficacy of concurrent chemotherapy with DC-CIK and CIK treatment in patients with treatment-refractory solid tumors.

Study treatment:

Patients in group A will receive 4 cycles of CIK treatments and 4 cycles of DC-CIK treatments within 8 months. Patients in group B will have no immunotherapy . chemotherapy are available in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with treatment-refractory advanced colorectal cancer can not accept operation .
2. Age 18 to 75 years.Eastern Cooperative Oncology Group (ECOG) score ≤ 2 points, estimate survival > 3 months;
3. Blood White Blood Cell(WBC)≥ 4×109/L, Hb ≥ 100g/L, Platelet Count(PLT)≥ 80×109/L; Alanine aminotransferase(ALT) and aspartate aminotransferase(AST)≤ 2 times of normal upper value; Serum Cr ≤ 2 normal upper value;
4. Without any other malignant disease;
5. With more than one scalable lesions
6. Patients Voluntary attempt, and informed consent.
7. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

Exclusion Criteria:

1. Patients who do not conform to the inclusion criteria;;
2. Patients with uncontrolled infection; underlying disease that was severe or life-threatening(such as uncontrolled brain metastasis ); Patients who were pregnant or lactating;
3. ECOG perform status ≥ 2;
4. Other situations that the researchers considered unsuitable for this study (such as mental illness, drug abuse, etc.)..

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, China

IPD SHARING:
Plan to Share IPD: Undecided